CLINICAL TRIAL: NCT06515301
Title: Key Interventions to Improve the Follow-up Adherence Post Cervical Precancerous Lesion Treatment in Ethiopia: A Pragmatic Randomized Controlled Trial
Brief Title: Key Interventions to Improve the Follow-up Adherence Post Cervical Precancerous Lesion Treatment in Ethiopia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Addis Ababa University (Other)
Responsible Party: Principal Investigator, Alemnew Destaw Mezgebu, Mr, Addis Ababa University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 008/24/SPH
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Suspicious Cervical Cancer Lesions Follow up Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Structured nurse-led telephone call reminders plus standard care. (Experimental): Participants in this arm will receive proactive telephone call reminders from nurses for their scheduled follow-up visits. Reminders will be administered initially at 4 months post-recruitment and then every 4 months for a year for HIV-negative women. For women living with HIV, reminders will be administered every 2 months for 6 months after recruitment.
  Interventions: Behavioral: Intervention 1: Structured nurse-led telephone call reminders. Intervention 2: Home-visit reminders by health extension workers. Intervention 3: Application-based automated SMS text reminders.
- Home-visit reminders by health extension workers plus standard care. (Experimental): Health Extension Workers (HEWs) will conduct home visits to remind participants of their scheduled follow-up appointments. Scheduled initially at 4 months post-recruitment for HIV-negative women and 2 months for HIV-positive women, followed by visits every 2 months for 6 months for HIV-positive individuals and every 4 months for 12 months for HIV-negative individuals.
  Interventions: Behavioral: Intervention 1: Structured nurse-led telephone call reminders. Intervention 2: Home-visit reminders by health extension workers. Intervention 3: Application-based automated SMS text reminders.
- Application-based automated SMS text reminders plus standard care. (Experimental): Participants will receive automated SMS text reminders via a mobile application for their follow-up visits. SMS reminders will be sent initially at 4 months and 2 months post-recruitment for HIV-negative and HIV-positive women, respectively. Subsequent reminders will be sent every 2 months for 6 months for HIV-positive women and every 4 months for 12 months for HIV-negative women.
  Interventions: Behavioral: Intervention 1: Structured nurse-led telephone call reminders. Intervention 2: Home-visit reminders by health extension workers. Intervention 3: Application-based automated SMS text reminders.
- Standard care only (Active Comparator): Participants in the control group will receive standard follow-up care according to the guidelines outlined by the Ethiopian Ministry of Health and current clinical practices of the country.These women will be orally informed of their follow-up appointment dates and will receive a post-treatment follow-up card at the baseline. Apart from this information and routine care, no additional interventions will be provided.
  Interventions: Behavioral: Intervention 1: Structured nurse-led telephone call reminders. Intervention 2: Home-visit reminders by health extension workers. Intervention 3: Application-based automated SMS text reminders.

INTERVENTIONS:
Behavioral: Intervention 1: Structured nurse-led telephone call reminders. Intervention 2: Home-visit reminders by health extension workers. Intervention 3: Application-based automated SMS text reminders. — Information already available

SUMMARY:
The goal of this pragmatic randomized control trial is to evaluate the effectiveness of three interventions in improving follow-up adherence among women treated for suspicious cervical lesions in primary healthcare settings in Ethiopia. The interventions include structured nurse-led telephone call reminders, home-visit reminders led by health extension workers, and application-based automated SMS text reminders. The main questions it aims to answer are:

* Does structured nurse-led telephone call reminders improve follow-up adherence among women treated for suspicious cervical lesions compared to standard care?
* Does home-reminder visits led by a Health Extension Worker (HEW) improve follow-up adherence among women treated for suspicious cervical lesions compared to standard care?
* Does app-based automated SMS reminders improve follow-up adherence among women treated for suspicious cervical lesions compared to standard care?

Structured Nurse-Led Telephone Call Reminders

* Participants will receive proactive phone call reminders for scheduled follow-up visits.
* The intervention includes three rounds: initially at 4 months post-recruitment, then every 4 months for HIV-negative women over a year, and every 2 months for 6 months for women living with HIV.

Home-Reminder Visits Led by HEW Health Extension Workers (HEWs) will conduct door-to-door visits to remind participants of their scheduled follow-up appointments.

• Door-to-door Visits will occur initially at 4 months (for HIV-negative women) and 2 months (for HIV-positive women) post-recruitment, then every 2 months for 6 months for HIV-positive and every 4 months for 12 months for HIV-negative participants.

App-Based Automated SMS Reminders

* Participants will receive SMS-based reminders for their follow-up visits.
* The intervention consists of three rounds: initial texts at 4 months and 2 months post-recruitment for HIV-negative and HIV-positive women, respectively, followed by reminders every 2 months for 6 months for HIV-positive women and every 4 months for 12 months for HIV-negative women.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 30-49 (HIV-negative).
* Women over 25 (HIV-positive).
* Treated for suspicious cervical lesions after a positive VIA screening.

Exclusion Criteria:

* History of hysterectomy.
* Diagnosis of other histological invasive cervical cancer.
* Suspicious cervical cancer cases.
* Pregnancy.
* Prior screening history.
* Vaginal bleeding.
* Lack of consent.

Ages: 25 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 466 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-11-20 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of adherence to follow up recommendations in the intervention and standard group after suspicious cervical cancer lesion treatment. | re-screening (VIA) after one year (11-13 months)
  Follow up adherence will be measured re-screening (VIA) after one year (11-13 months after first screening). We will use objective measurement thorough review of the comprehensive records maintained within the cervical cancer screening follow-up registry.Accordingly, women who fail to return for their scheduled follow-up visit will be categorized as "Lost to Follow-Up", while those who do attend will be categorized as "Follow-Up Adherent

CONTACTS AND LOCATIONS:
Locations (1):
- Worabe Health Center, Silte, Southern Ethiopia, Ethiopia

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared to maintain participant confidentiality and comply with ethical guidelines. However, aggregated, de-identified data will be made available upon reasonable request after study completion and publication. Requests should be directed to the corresponding author, and data access will be provided in line with institutional policies and BMJ Open's data-sharing policy requirements.

REFERENCES:
- [Derived] Destaw A, Getachew S, Getachew E, Shita A, Midaksa M, Rossner SS, Kroeber ES, Addissie A, Kantelhardt EJ, Gizaw M. Follow-up rescreening uptake and persistent positive rates among women after positive cervical cancer screening results in Ethiopia: a longitudinal cross-sectional study. BMJ Open. 2025 Jul 28;15(7):e099955. doi: 10.1136/bmjopen-2025-099955. PMID 40730399
- [Derived] Destaw A, Getachew S, Getachew E, Shita A, Midaksa M, Rossner S, Kroeber ES, Addissie A, Kantelhardt EJ, Gizaw M. Study protocol for key interventions to improve the follow-up adherence postcervical precancerous lesion treatment in Ethiopia: a pragmatic randomised controlled trial. BMJ Open. 2025 Jan 7;15(1):e091693. doi: 10.1136/bmjopen-2024-091693. PMID 39773801